CLINICAL TRIAL: NCT01684046
Title: Evaluation of the Effectiveness of Two Marketed Multi-Purpose Solutions for Silicone Hydrogel Contact Lenses - Study 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: M-12-041
Record Dates: First submitted 2012-09-10; First posted 2012-09-12 (Estimated); Results first posted 2014-04-29 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-03

CONDITIONS: Myopia; Hyperopia; Contact Lens Comfort
Keywords: multi-purpose solution; silicone hydrogel; contact lenses; comfort; Opti-Free; RevitaLens
MeSH Terms: conditions — Myopia; Hyperopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PureMoist - RevitaLens (Other): Opti-Free® PureMoist® MPDS used first, followed by RevitaLens MPDS. Each product used as indicated for 30 days with participant's habitual contact lenses.
  Interventions: Device: Opti-Free® PureMoist® MPDS; Device: RevitaLens MPDS; Device: Habitual Contact Lenses
- RevitaLens - PureMoist (Other): RevitaLens MPDS used first, followed by Opti-Free® PureMoist® MPDS. Each product used as indicated for 30 days with participant's habitual contact lenses.
  Interventions: Device: Opti-Free® PureMoist® MPDS; Device: RevitaLens MPDS; Device: Habitual Contact Lenses

INTERVENTIONS:
Device: Opti-Free® PureMoist® MPDS
  Other Names: OPTI-FREE® PureMoist®
Device: RevitaLens MPDS
  Other Names: RevitaLens OcuTec®; COMPLETE® RevitaLens
Device: Habitual Contact Lenses — Silicone hydrogel contact lenses per participant's habitual brand, prescription, and replacement schedule worn on a daily wear basis for at least 8 hours a day, 5 days a week for the duration of the study. During the washout period, the contact lenses were worn on a daily disposable basis.

SUMMARY:
The purpose of this study was to evaluate the performance of Opti-Free® PureMoist® Multi-purpose Disinfecting Solution (MPDS) compared to AMO RevitaLens OcuTec® MPDS (US brand name)/COMPLETE RevitaLens (Europe brand name) in silicone hydrogel contact lens wearers.

DETAILED DESCRIPTION:
In this 2-period crossover study, eligible participants were randomized to either Opti-Free® PureMoist MPDS or RevitaLens MPDS in Period 1 for use with their habitual contact lenses, after which they switched to the alternate solution in Period 2. Each period was 30 days in length. A 2-day washout period during which participants refrained from using a multi-purpose contact lens solution preceded Period 1 and Period 2.

ELIGIBILITY:
Inclusion Criteria:

* Wear single vision sphere silicone hydrogel contact lenses (CooperVision™ Biofinity®, Alcon® Air Optix® Aqua, Bausch+Lomb® PureVision™ or ACUVUE® Oasys™) on a daily wear basis (a minimum of 8 hours per day, 5 days a week) for at least 1 month prior to Visit 1;
* Willing to wear lenses on a daily wear basis (a minimum of 8 hours per day, 5 days a week) for the duration of the study, and wear lenses for 16 hours on 2 days during the study;
* Must have habitually used a biguanide preserved multi-purpose solution (other than RevitaLens) for at least 30 days prior to Visit 1;
* Vision correctable to 20/30 Snellen (feet) or better in each eye at distance with pre-study contact lenses at Visit 1;
* Have access, capability and willingness to review and answer text messages;
* Read, sign, and date IRB/IEC approved informed consent and privacy document before enrollment;
* Willing to follow the study procedures and visit schedule;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Need to wear lenses on an extended wear (i.e overnight) basis during the study;
* Known sensitivity or intolerance to biguanide, polyquaternium-1 (POLYQUAD), or ALDOX preserved lens care products;
* Monocular (only one eye with functional vision) or fit with only one lens;
* Wearing toric or multifocal contact lenses or fit with monovision;
* Use of additional lens care products other than a biguanide preserved multi-purpose solution such as daily or enzyme cleaners within the 1 week prior to Visit 1;
* Use of topical ocular over-the-counter (OTC) or prescribed topical ocular medications, with the exception of rewetting drops, within 7 days prior to Visit 1;
* Abnormal ocular condition observed during the Visit 1 slit-lamp examination;
* Current or history of ocular infections or severe inflammation within 6 months prior to Visit 1;
* Ocular surgery within the 12 months prior to Visit 1;
* Participation in any other clinical trial within 30 days of enrollment;
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2012-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessie Lemp, MS, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 5 study centers located in the US, 2 study centers located in the UK, and 3 study centers located in Germany.
Pre-assignment Details: Of the 196 enrolled, 4 participants were exited as screen failures prior to randomization. This reporting group includes all randomized participants who were exposed to a study regimen (test or control) (192).
Groups:
- PureMoist - RevitaLens: Opti-Free® PureMoist® MPDS, followed by RevitaLens MPDS. Each product used as indicated for 30 days with participant's habitual contact lenses.
- RevitaLens - PureMoist: RevitaLens MPDS, followed by Opti-Free® PureMoist® MPDS. Each product used as indicated for 30 days with participant's habitual contact lenses.
Period: Period 1, First 30 Days
Arm/Group | PureMoist - RevitaLens | RevitaLens - PureMoist
Started | 97 | 95
Completed | 97 | 93
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 2
Period: Period 2, Second 30 Days
Arm/Group | PureMoist - RevitaLens | RevitaLens - PureMoist
Started | 97 | 93
Completed | 97 | 93
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all participants who were exposed to a study regimen (test or control).
Groups:
- PureMoist / RevitaLens: Opti-Free® PureMoist® MPDS and RevitaLens MPDS used during Period 1 and Period 2 in randomized order in crossover assignment.
Arm/Group | PureMoist / RevitaLens
Number analyzed (Participants) | 192
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.0 (11.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 142
  Male | 50

OUTCOME MEASURES:

1. Primary Outcome: Subjective Lens Wear Comfort
Description: Lens wear comfort was assessed by the participant on a 5-point Likert scale. The participant was instructed to select a single response to the statement, "When I use this solution, I can comfortably wear my lenses," with 1 = strongly disagree, 2 = disagree, 3 = neither agree nor disagree, 4 = agree, and 5 = strongly agree.
Time Frame: Day 30
Population: This analysis population includes all participants who were exposed to study regimen (test and control) and completed both study periods, excluding major protocol deviations.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- PureMoist: Opti-Free® PureMoist® MPDS used during Period 1 or Period 2 for 30 days with participant's habitual contact lenses.
- RevitaLens: RevitaLens MPDS used during Period 1 or Period 2 for 30 days with participant's habitual contact lenses.
Arm/Group | PureMoist | RevitaLens
Number analyzed (Participants) | 183 | 183
units on a scale | 4.3 (0.89) | 4.3 (0.72)

ADVERSE EVENTS:
Time Frame: Adverse events (AE) were collected for the duration of the study (4 months). AEs were elicited by non-direct questioning of the participant and spontaneous reporting by the participant. AEs were recorded at every visit.
Description: An AE was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs in subjects, users or other persons, whether or not related to the medical device. This analysis population includes all participants who were exposed to a study regimen (test or control), based on treatment-specific exposure.
Arm/Group | PureMoist | RevitaLens
Serious Adverse Events (participants affected / at risk) | 0/190 | 0/192
Other Adverse Events (participants affected / at risk) | 0/190 | 0/192

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.